CLINICAL TRIAL: NCT02694757
Title: Pilot Study to Evaluate the Efficacy of Ostom-i Alert System at Decreasing Dehydration Related Complications in Patients With New Ileostomies
Brief Title: Efficacy of Ostom-i Alert System at Decreasing Dehydration Related Complications
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Liliana Bordeianou, Associate Professor of Surgery, Division of General and Gastrointestinal Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGH2015-P-000873
Record Dates: First submitted 2016-02-25; First posted 2016-02-29 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Ileostomy - Stoma
Keywords: Ostom-i; OIA device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ostom-i device (Experimental): Subjects will receive an Ostom-i device which will be worn over the ostomy bag underneath the subject's clothing. Output will be monitored daily by the Ostom-i application.
  Interventions: Device: Ostom-i device

INTERVENTIONS:
Device: Ostom-i device — The Ostom-i alert (OIA) is a discrete novel device which clips onto any ostomy bag from edge to edge and measures the horizontal tension between the edges over time, as a result of stool volume in the ostomy. It is an FDA approved medical device.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Ostom-i device in decreasing readmission rates of subjects with new ileostomies in the first 30 days post-operatively.

DETAILED DESCRIPTION:
Ileostomy creation is a common surgery performed in patients who have disease or injury to their colon requiring fecal diversion. Ileostomy formation can be temporary, and is often used to protect anastomoses in colorectal resections. It can also be permanent, when disease or injury is more extensive. All patients undergoing an ileostomy face unique post-operative challenges due to the alteration of absorption and waste elimination pathways. Prior to surgery, patients are counseled about these challenges including the expected increase in frequency of liquid stools, which can have both bothersome and more serious complications.

Hospital readmissions in people who have recently undergone colon and rectal surgery are frequent, and can be costly and delay post-operative healing . Current NSQIP colectomy readmission rates for open and laparoscopic colectomies over the past 12 months at Massachusetts General Hospital were 11.3% and 10.9% respectively. Average national readmission rates for open and laparoscopic colectomies over the past 12 months were 13.2% and 10.7% respectively. The most common reason for hospital readmission following surgery is dehydration, with other causes including infection, bowel obstruction, bleeding, wound dehiscence with leak, and pain.

Dehydration is a serious but preventable complication in patients with new ileostomies. Even small changes in fluid intake or output can cause body fluid imbalances that promote dehydration and necessitate IV rehydration . Previous research has shown that the use of pre-operative teaching, direct patient engagement from post-op day one, engaging patients to perform self-care for their stoma during hospitalization, and having patients track intake and output post-discharge can decrease readmission rates . With implementation of this pathway over the course of 7 months, there was a decrease in the overall 30- day postdischarge readmission rate for patients with new ileostomies from 35.4% to 21.4%, with the rate for dehydration alone falling from 15.5% to 0% .

The Ostom-i alert (OIA) is a discrete novel device which clips onto any ostomy bag from edge to edge and measures the horizontal tension between the edges over time, as a result of stool volume in the ostomy. It is an FDA approved medical device.

Until now, the OIA has been mainly used to warn patients when the ostomy bag is at risk of overflow thereby reducing the risk of leakage causing embarrassment to the patient and caregivers. It can also be used to evaluate the overall output of the ostomy. When patients leave the hospital, the OIA data is sent to the patient's smartphone through bluetooth technology and can be viewed on the internet in real time by the surgical team (stoma nurse, surgeon, clinical research staff). This would allow patients to monitor their output more accurately and allow them to contact clinical staff with questions or to help with bowel management when output is outside of established parameters (too little or too high output).

While all patients with ileostomy have a risk of dehydration, early identification of those at greater risk may lead to home intervention and decreasing hospital readmission. Decreased readmissions ultimately leads to faster post-operative recovery, decreased risk of sequela of readmission (nosocomial infection, pneumonia etc) and decreased healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* English speaking
* creation of new ileostomy
* access to smartphone with bluetooth technology to support OIA application
* able to give written consent
* have preoperative counseling about stoma with ostomy nurse (excludes emergent ostomy creation)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Bordeianou, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messaris E, Sehgal R, Deiling S, Koltun WA, Stewart D, McKenna K, Poritz LS. Dehydration is the most common indication for readmission after diverting ileostomy creation. Dis Colon Rectum. 2012 Feb;55(2):175-80. doi: 10.1097/DCR.0b013e31823d0ec5. PMID 22228161
- [Background] Nagle D, Pare T, Keenan E, Marcet K, Tizio S, Poylin V. Ileostomy pathway virtually eliminates readmissions for dehydration in new ostomates. Dis Colon Rectum. 2012 Dec;55(12):1266-72. doi: 10.1097/DCR.0b013e31827080c1. PMID 23135585

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ostom-i Device
Started | 3
Completed | 0
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: Because none of the study participant completed the study, there are no participant data to anaylze
Arm/Group | Ostom-i Device
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39 [23 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Readmission Rate
Description: No outcomes were measured due to termination of study.
Time Frame: 30 days post-operation
Population: No analysis was completed due to termination of study.
Arm/Group | Ostom-i Device
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ostom-i Device
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT02694757/Prot_SAP_000.pdf